CLINICAL TRIAL: NCT02755337
Title: The Evaluation of Lung Cancer Patient Treated With Epidermal Growth Factor Receptor Tyrosine Kinase
Acronym: EVALUATE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Soetomo General Hospital (Other Government)
Responsible Party: Principal Investigator, Laksmi Wulandari, MD, PhD, FCCP, MD, PhD, Dr. Soetomo General Hospital
Other Study IDs: Dr. Soetomo General Hospital
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: adenocarcinoma; non-adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate Non-Small Cell Lung Cancer (NSCLC) patients clinical profile and the outcome after treatment with Gefitinib in Pulmonary Oncology Outpatient Clinic Dr. Soetomo General Hospital, Surabaya, Indonesia.

DETAILED DESCRIPTION:
Primary Objective: To determine the efficacy of Gefitinib in NSCLC patient harboring a positive EGFR mutation.

Secondary Objective: To evaluate the subjective response of NSCLC patients harboring a positive EGFR mutation who treated with Gefitinib.

Safety Objective: To evaluate the safety and tolerability of Gefitinib in NSCLC patient harboring a positive EGFR mutation.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC based on histopathologic examination
* Adenocarcinoma and/or nonadenocarcinoma based on histology examination
* Clinical stadium stage IIIB and IV
* Age 16-70 years old
* Received gefitinib as therapy
* At least completed 2 (two) data sets of RECIST 1.1 evaluations during the study period from January 2013 until July 2015

Exclusion Criteria:

* Missing data of any variables of the treatment outcomes in the medical record

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: NSCLC patients (adenocarcinoma and non-adenocarcinoma histology) who harbor a positive EGFR mutation and receive Gefitinib (Iressa) as treatment.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
PFS (Progression Free Survival) | through study completion, in average of 1 year
  Progression Free Survival (PFS) as defined by RECIST 1.1 or attending physician's clinical judgement of clinical progression state
Overall Survival (OS) | through study completion, in average of 1 year
  Overall Survival (OS) as defined by the date of death certificate given by the attending physician or by other government officials

CONTACTS AND LOCATIONS:
Overall Officials: Laksmi Wulandari, MD, PhD, Principal Investigator — Dr. Soetomo General Hospital
Locations (1):
- Dr. Soetomo General Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No